CLINICAL TRIAL: NCT01393483
Title: A Prospective Clinical Trial to Evaluate Mesothelin as a Biomarker for the Clinical Management of Esophageal Adenocarcinoma (EAC)
Brief Title: Evaluate Mesothelin as a Biomarker for the Clinical Management of Esophageal Adenocarcinoma (EAC)
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 11-037
Record Dates: First submitted 2011-07-11; First posted 2011-07-13 (Estimated); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Esophageal Cancer; Adenocarcinoma
Keywords: esophagectomy; endoscopy; biopsy; Tissue mesothelin; Serum mesothelin; 11-037
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — tissue and serum

GROUPS / COHORTS (3):
- patients endoscopically resected: In patients with endoscopically resected T1 disease (40 patients in 2 years) if available, we will stain the initial endoscopic tumor specimen, as well as any subsequent specimen obtained at each routine 3(+/- 2) month interval endoscopy.
  Interventions: Other: serum and tissue mesothelin
- patients treated primarily with surgery: In patients who undergo surgery as their primary therapy, serum will be obtained at the time of surgical resection, and at each subsequent long-term disease status follow-up visit every 4 (+/- 2) months.
  Interventions: Other: serum and tissue mesothelin
- patients who undergo chemo-radiation prior to surgery: a serum sample will be obtained : 1) prior to initiation of therapy, 2) following the completion of induction chemotherapy, 3) at the time of surgical resection, and 4) at each subsequent long-term disease status follow-up visit every 4 (+/- 2) months. The availability of tissue for staining will determine whether or not patients are evaluable for Group 3.
  Interventions: Other: serum and tissue mesothelin

INTERVENTIONS:
Other: serum and tissue mesothelin — Tissue mesothelin staining at the time of the initial endoscopy, and of any subsequent biopsy specimen during the endoscopic screening period.
  Serum mesothelin level at the time of initial endoscopy, and at each subsequent endoscopy for two years or until disease recurs.
  Groups: patients endoscopically resected
Other: serum and tissue mesothelin — Tissue mesothelin staining on the surgically resected esophageal specimen. Serum mesothelin level at the time of surgical resection, and at each follow-up clinic visit for two years or until disease recurs.
  Groups: patients treated primarily with surgery
Other: serum and tissue mesothelin — Tissue mesothelin staining on the initial endoscopic specimen (typically obtained when an EUS is done) and on the surgically resected esophageal specimen Serum mesothelin level prior to initiation of induction chemotherapy, at the time of the post-induction PET, at the time of surgical resection, and at each follow-up clinic visit for two years or until disease recurs.
  Groups: patients who undergo chemo-radiation prior to surgery

SUMMARY:
The purpose of this study is to find out whether a protein, called mesothelin, found in the blood and tissue can be used as "marker" for esophageal cancer. Doctors at Memorial Sloan-Kettering Cancer Center would like to compare levels of this protein in patients with abnormal cells or tissue of the esophageal to the levels of this protein in patients being treated for cancer for the esophagus.

ELIGIBILITY:
Inclusion Criteria:

* Patients with T1 adenocarcinoma or suspected adenocarcinoma who are scheduled for a biopsy and mucosal resection (Group 1)
* Patients with a T1-2N0 adenocarcinoma or suspected adenocarcinoma who are scheduled to undergo and esophagectomy (Group 2)
* Patients with T2N1 and T3N0-1 adenocarcinoma or suspected adenocarcinoma who are scheduled to undergo endoscopy and biopsy and/or endoscopic ultrasound and biopsy prior to pre-operative chemo-radiotherapy and have baseline and surgical tissue available for staining (Group 3)

Exclusion Criteria:

* Patients <18 years of age
* Patients unfit medically for endoscopy surveillance and therapy
* Patients unfit medically for esophagectomy
* Patients with stage IV esophageal adenocarcinoma
* Patients previously treated with chemo-radiotherapy for their esophageal cancer
* Patients with squamous cell carcinoma of the esophagus
* Patients who have a history of cancer within 3 years or have a concurrent cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient seen in the gastroenterology and thoracic clinics who fits the inclusion criteria will be approached by the treating physician, the protocol investigator, or thoracic research team at Memorial Sloan-Kettering Cancer Center (MSKCC
Sampling Method: Non-Probability Sample
Enrollment: 371 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-10-22 (Actual)

PRIMARY OUTCOMES:
To evaluate prospectively what proportion of esophageal adenocarcinomas express tissue. | 2 years
  The investigators will examine the range and variability in the percentage on cells stained (for TM) and in the absolute value (for SM). TM expression is commonly analyzed in a binary fashion, with 25% of cells stained indicating positive expression (per standard pathological guidelines for tissue staining)
To evaluate prospectively if serum mesothelin levels correlate to clinical stage in esophageal adenocarcinomas | 2 years
  The investigators will explore the optimal cut point that defines positive expression. Serum mesothelin (SM) will be measured and analyzed whenever possible on a continuous scale.
To evaluate prospectively if clinical response to induction chemotherapy | 2 years
  First, the investigators will use two-sample t-tests to determine whether the initial responders to induction chemotherapy (defined as >30% decrease in SUV at the repeat PET) differ from non-responders in their 1) baseline (pre-induction) SM value, and 2) percent change in SM value between pre-induction and mid-induction (after 2 cycles) evaluations.
To evaluate prospectively if clinical response to concurrent chemo-radiation correlates to serum mesothelin levels | 2 years
  The investigators will take the following steps in order to assess the ability of SM at the time of resection with curative intent to predict disease recurrence: 1) we will examine the association between SM and the risk of recurrence by fitting a Cox proportional hazards model (after appropriate transformation of the SM value and checking of the PH assumption

SECONDARY OUTCOMES:
To evaluate whether expression of tissue mesothelin is a predictor of recurrence | 2 years
  The investigators will Wilcoxon test to investigate the association between serum mesothelin and tissue mesothelin at each time point where both markers are evaluated, and will further attempt to obtain an aggregate measure of this correlation using clustered Wilcoxon test, which accounts for multiple measurements per patient (14).
To evaluate whether expression of tissue mesothelin is a predictor of poor response to chemotherapy | 2 years
  Mesothelin positive tumors (MES+) will be defined as strong staining in > 25% of the tumor cells and mesothelin negative tumors (MES-) are defined as <= 25% cytoplasmic staining. Serum mesothelin will be collected and analyzed, whenever possible, on a continuous scale.
To evaluate for the presence of any confounders in the putative association between serum mesothelin expression and the risk of recurrence | 2 years
To evaluate the correlation between serum mesothelin levels and tissue expression | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Prasad Adusumilli, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Rizk NP, Servais EL, Tang LH, Sima CS, Gerdes H, Fleisher M, Rusch VW, Adusumilli PS. Tissue and serum mesothelin are potential markers of neoplastic progression in Barrett's associated esophageal adenocarcinoma. Cancer Epidemiol Biomarkers Prev. 2012 Mar;21(3):482-6. doi: 10.1158/1055-9965.EPI-11-0993. Epub 2012 Jan 11. PMID 22237988
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm